CLINICAL TRIAL: NCT06893965
Title: Intra Ocular Pressure Monitoring After Intravitreal Injection of Aflibercept 8mg/0.07mL
Brief Title: Acute Intra Ocular Pressure Monitoring After Aflibercept 8mg/0.07mL
Acronym: AFLIPIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Sainte-Anne Military Teaching Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-CHITS-001; 2025-A00113-46 (Other: ID-RCB number)
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Macular Diseases
Keywords: Diabetic Macula Edema; Intravitreal injection; Anti-VEGF; Aflibercept; Wet age-related macular degeneration (AMD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOP Monitoring (Other)
  Interventions: Diagnostic Test: Intra ocular pressure Measure

INTERVENTIONS:
Diagnostic Test: Intra ocular pressure Measure — Measurement of IOP before injection (T0), just after the injection (T1) then 15 (T15), 30 (T30) and 45 (T45) minutes after the injection. Measurement are done with Perkins Tonometer

SUMMARY:
In just a few years, intravitreal injections have become a standard method of administration for certain retinal deseases (age-related macular degeneration [AMD], diabetic edematous maculopathy or retinal vein occlusion [RVO]). Thus, vascular endothelial growth factor (anti-VEGF) inhibitors are injected repetitively, every 4 to 6 weeks, in some patients in order to treat such pathologies.

It is established that each of these IVTs has repercussions on the intraocular pressure (IOP) of patients. They immediately present with an intraocular pressure spike (IOP reaching nearly 50mmHg) for a duration of a few minutes (between 15 and 30 minutes) when the injected volume is 0.05mL, which is currently used.

In order to reduce the frequency of injections in patients, higher concentrations of active ingredients with anti-VEGF properties will arrive on the market with higher injection volumes of up to 0.07mL (marketing of Aflibercept 8mg/0.07ml in France since 01/06/2025. As IOP spikes are linked to the volume injected, the repercussions of such volumes could probably be greater and require additional actions. Indeed, currently the volumes used (0.05mL) rarely lead to complications such as transient blindness secondary to ocular hypertonia. In this case, an anterior chamber puncture may be necessary.

To date, the impact on IOP of the 0.07mL injection has not yet been evaluated in the short and long term. Indeed, the repetition of IVT leads to a repetition of IOP peaks of around 50mmHg in the same patient. Some studies have analyzed the anatomical repercussions on the optic nerve of these peaks and have noted a reduction in the thickness of the peripapillary nerve fibers (RNFL for Retinal Nerve Fiber Layer) in Optical Coherence Tomography (OCT for Optical Coherence Tomography) after the 3 monthly IVTs recommended for the induction phase of treatment. But other studies have not found a significant drop in RNFL after several years of regular treatment with IVT. The studies were all carried out with volumes of 0.05mL and the repercussions with a volume of 0.07mL are therefore not reported in the literature.

The AFLIPIO study aims to study the short-term pressure profile after performing an IVT of Aflibercept, at a volume of 0.07mL, and to evaluate the longer-term anatomical repercussions (12 months) on the head of the optic nerve when repeating IVT of Aflibercept, at a volume of 0.07mL.

DETAILED DESCRIPTION:
In order to reduce the frequency of injections in the so-called sub-optimal patients, a "new generation" anti-VEGF will arrive on the market with higher concentrations of active ingredients with a higher injection volume of 0.07mL (marketing of Aflibercept 8mg/0.07ml in France since 01/06/2025). As IOP peaks are linked to the volume injected, the repercussions of such volumes could probably be higher and require additional procedures. In fact, currently the volumes used (0.05mL) rarely lead to complications such as transient blindness secondary to ocular hypertonia. In this case, an anterior chamber puncture may be necessary. To date, the pressure profile after IVT of 0.07mL is not known, on experimental ocular models, the IOP after an IVT of 0.07mL could reach more than 70mmHg with a return to normal after 20 to 25 minutes. So to evaluate the IOP profile after intravitreal injection of Aflibercept 8mg/0.07mL, the IOP will be monitored after an injection during 45 minutes. IOP will be measure with a Perkins Tonometer in order to have aplanation results. Measures will be done just before and after the injection and at 15minutes, 30 minutes and 45 minutes.

To evaluate the risk of transient monocular blindness, we will note all transient blindness after the injection.

The longer-term repercussions are also not known. Indeed, the repetition of IVT leads to a repetition of IOP peaks in the same patient. The previous studies were all carried out with volumes of 0.05mL and the repercussions with a volume of 0.07mL are therefore not reported in the literature and deserve to be researched. In order to evaluate the repercussion of the new volume, Retinal Nerve Fiber Layer assessed with Optical Coherence tomography will be done just before the injection and at the end of the follow up 12 months +/-2 months.

The treatment regimen will not be modified by the study.

The inclusion visit will be carried out during a routine care consultation. During this consultation, patients will be informed of the research and will be included once their consent has been obtained. The patient's inclusion can take place during the first IVT or during another IVT of the patient's follow-up.

During this visit, the investigator will carry out:

* A papillary OCT before IVT. This is a non-invasive light imaging technique which makes it possible to obtain cross-sectional images of the papilla and to evaluate in particular the therapeutic response to IVT,
* A first measurement of the IOP before injection (T0) by a PERKINS applanation tonometer. It uses an applanation tonometry technique, namely the measurement of IOP by counter pressure on the cornea, after the instillation of anesthetic eye drops.
* Then, injection of Aflibercept 8mg/0.07mL following the usual recommendations of the service,
* and new IOP measurements just after the injection (T1) then at 15 (T15), 30 (T30) and 45 (T45) minutes after the injection.

The consultation will therefore be extended by an additional 45 minutes compared to a traditional consultation. The application of a local anesthetic will also be added by the research to carry out IOP measurements at 30 and 45 minutes (the previous measurements, ie. T1 and T15, will benefit from the local anesthesia of the IVT carried out for current practice).

At the end of this consultation, there will be no change in patient monitoring in terms of frequency of consultations and subsequent injections. IOP measurements will only be taken during the first inclusion consultation.

Patients will perform a new papillary OCT 1 year after the injection where the IOP was monitored, i.e. 1 year after inclusion in the research.

Follow-up for research will end after the papillary OCT at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over;
* Patient with an indication for Aflibercept 8mg/0.07mL (EYLEA 8mg)
* Naive or switched patient, i.e. so-called suboptimal responder to anti-VEGF with high injection frequencies
* Patient with rights to social security
* Having given free and informed consent before any participation in research.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under legal protection (guardianship, curatorship, etc.) or legal protection
* Patient with significant astigmatism distorting the IOP values in applanation
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular Pressure | At baseline : just before injection (T0), just after injection (T1) and at 15 minutes (T15), 30 minutes (T30) and 45 minutes after injection (T45)
  Measurement performed with Perkins Tonometer, results in mmHg

SECONDARY OUTCOMES:
Retinal Nerve Fiber Layer (RNFL) | At baseline before the intravitreal injection (T0) and 1 year
  RNFL will be assessed using Optical Coherence Tomography (OCT) before the first injection of the study (T0) and at one year of patient follow-up (M12): measurement of the RNFL (Retinal Nerve Fiber Layer or thickness of the peripapillary nerve fibers).
Number of patients who experienced transient monocular blindness | In the minute following intravitreal injection
  Evaluation the hand motion after the intravitreal injection
IOP evolution in the glaucoma patient subgroup | At baseline : just before injection (T0), just after injection (T1) and at 15 minutes (T15), 30 minutes (T30) and 45 minutes after injection (T45)
  Changes in intraocular pressure will be assessed in a specific subgroup of patients treated for glaucoma.

CONTACTS AND LOCATIONS:
Overall Officials: Hussam EL CHEHAB, MD, FEBO, Study Director — Military Hospital of Sainte Anne, Toulon, France
Locations (1):
- Military Hopsital of Sainte Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No